









## **CONSENT FORM**

**Title of Project**: Developing an intervention to help nurses improve the assessment and care of the sexual health needs of men with Inflammatory Bowel Disease: a mixed methods study using coproduction (MenSH-IBD)

| <b>IRAS ID:</b> 334340 | | Participant Number |
|---|---|---|
| | ad the opportunity to | Pleas initial behave the information, ask questions and have had |
| 2. I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my legal rights being affected. I understand any information collected until the point of withdrawal will be included in the study. | | |
| 3. I understand that the information I provide will be used to support other research in the future and may be shared anonymously with other researchers. | | |
| audio recorded so that<br>transcription service t | at they can be transcr<br>bound by a confidenti<br>sed but transcriptions | -production workshops (delete as appropriate) being ribed by a researcher or through a professional iality agreement. Recordings will be deleted when the (where identifiable information has been redacted) will |
| at the University of You | ork and York St John | y contact details may also be shared with researchers University who are supporting the administration of urely and only used for the purpose of this research. |
| 6. I understand that if the researcher thinks that I or someone else may be at risk of harm they will have to contact the relevant authorities. | | |
| 7. I agree to take part in the above study. | | |
| <ul> <li>OPTIONAL</li> <li>8. I give permission for my contact information to be held and maintained by York and Scarborough Teaching Hospitals NHS Foundation Trust to inform me of the study results and/or invite me to participate in future research studies for a maximum of 3 years following the end of the study.</li> </ul> | | |
| Name of Participant | Date | Signature |
| Name of Person | Date | Signature |

seeking consent